CLINICAL TRIAL: NCT06333587
Title: Multicenter International Prospective Analysis on Minimally Invasive Treatments of the Thyroid (MIPA- MITT) of of Micropapillary Thyroid Carcinoma
Brief Title: Minimally Invasive Treatments of the Thyroid
Acronym: MIPA-MITT
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1810
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Papillary Thyroid Microcarcinoma
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- image-guided thermal ablation: image-guided thermal ablation in patients with diagnosis of micropapillary thyroid carcinoma
  Interventions: Procedure: image-guided thermal ablation

INTERVENTIONS:
Procedure: image-guided thermal ablation — image-guided thermal ablation in patients with diagnosis of micropapillary thyroid carcinoma

SUMMARY:
This is a prospective cohort study to test Minimally Invasive Treatments of the Thyroid (MITT) as potential alternative to surgery in patients with Papillary Thyroid MicroCarcinoma (PTMC)

DETAILED DESCRIPTION:
Image-guided thermal ablations have been successfully applied in the treatment of several type of tumors, and have been recently proposed as a potential alternative to surgery also in patients with thyroid diseases, and named "Minimally Invasive Treatments of the Thyroid (MITT)". These minimally invasive treatments, compared to surgical treatment have similar efficacy, fewer complications, better quality of life, and better cosmetic outcomes. These procedures allow precise delivery of the heat locally to the lesion, sparing the surrounding thyroid tissue, and thus minimizing the invasiveness of the treatment and the impact on thyroid function.

This study aim to establish a prospective registry of the cases of patients treated with MITT for a Papillary Thyroid MicroCarcinoma (PTMC), in order to validate the safety of the procedure and to set the basis for collecting long term results in a large cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18years
* Patients with diagnosis of papillary thyroid microcarcinoma, citologically proven, suitable for MITT.
* Written informed consent must be signed and dated by the patient and the investigator prior to inclusion.
* Patients must be accessible for follow-up

Exclusion Criteria:

* Tumors > 1 cm, other citological type, refusal of MITT, unsuitable for MITT, unmanageable coagulative disorders
* Patients with psychiatric, addictive, or any disorder, which compromises ability to give informed consent for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid diseases suitable for "Minimally Invasive Treatments of the Thyroid (MITT)" as potential alternative to surgery
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with major complications occurring within one month after the date of intervention | 1 month
  Complications will be reported according to modified Society of Interventional Radiology (SIR) classification

SECONDARY OUTCOMES:
Percentage of patients with local recurrence at 10 years | 10 years
  Evaluation of disease free survival (DFS): percentage of patient whith a local recurrence at 10 years of follow up
Percentage of patients with distant metastasis at 10 years | 10 years
  Evaluation of disease free survival (DFS): percentage of patient whith distant metastasis at 10 years of follow up
Percentage of patients died at 10 years | 10 years
  Evaluation of Overall Survival (OS): Percentage of patients died at 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Mauri, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy